CLINICAL TRIAL: NCT05080231
Title: Blood Specimen Collection for COVID-19 Immunity Assessment Mailer Kit Clinical Study
Brief Title: COVID-19 Immunity Assessment
Status: Completed | Type: Observational
Sponsor: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT-0239
Record Dates: First submitted 2021-10-13; First posted 2021-10-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- COVID-19 Vaccinated Individuals: Males and females, 13years old and above, vaccinated for COVID-19
- Previously positive for COVID-19 and unvaccinated individuals: Males and females, 13years old and above, unvaccinated for COVID-19 and previously tested positive for COVID-19.
- No previous COVID infection or vaccination: Males and females, 13years old and above, unvaccinated for COVID-19 and previously not tested positive for COVID-19.

SUMMARY:
The purpose of this study is to collect blood specimens from individuals post infection or post vaccination over time to assess COVID19 Immunity.

DETAILED DESCRIPTION:
The DxTerity COVID-19 Immunity Assessment Collection Mailer Kit contains the DxCollect MicroCollection Device (MCD) Serology fingerstick blood collection device packaged as a home collection kit, designed for collection and shipment of fingerstick blood back to DxTerity CLIA (Clinical Laboratory Improvements Amendment) certified laboratory for testing.

The clinical performance of the collection device for use with anti-SARS-CoV-2 antibody tests will be evaluated for use with cPASS™ anti-SARS-CoV-2 neutralizing antibody detection kit (EUA 201427).

The samples may also be used for assessing immunity or protection post COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥13 years old.
* Not vaccinated and were previously positive for COVID-19 OR are vaccinated for COVID-19.
* Provides test report to demonstrate prior COVID-19 positive result (only applicable to unvaccinated subjects who were previously positive for COVID-19, not applicable for COVID-19 vaccinated subjects).
* Provides informed consent and completed questionnaire.
* Able to register the collection kit on the DxTerity portal.
* Able to collect and ship blood samples back to DxTerity.

Exclusion Criteria:

* Unable to provide COVID-19 positive test report (only applicable to unvaccinated subjects who were previously positive for COVID-19, not applicable for COVID-19 vaccinated subjects).
* Unable to complete informed consent and/or questionnaire.
* Unable to complete the study activities in a timely manner.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Males and females ≥13 years old. Not vaccinated and were previously positive for COVID-19 OR are vaccinated for COVID-19.
  Provides test report to demonstrate prior COVID-19 positive result (only applicable to unvaccinated subjects who were previously positive for COVID-19, not applicable for COVID-19 vaccinated subjects).
  Provides informed consent and completed questionnaire. Able to register the collection kit on the DxTerity portal. Able to collect and ship blood samples back to DxTerity.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Neutralizing Antibody Levels | 3 months
  Measuring neutralizing antibody levels with COVID-19 immunity assessment test

CONTACTS AND LOCATIONS:
Locations (1):
- DxTerity Diagnostics Inc., Compton, California, United States